CLINICAL TRIAL: NCT02044939
Title: Pulmonary Rehabilitation in Fibrotic Pulmonary Sarcoidosis (Stage IV): Randomized Controlled Trial
Brief Title: Pulmonary Rehabilitation in Patients With Sarcoidosis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough recruitment
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011_23/1917; 2012-A00347-36 (Other: ID-RCB Number, ANSM)
Record Dates: First submitted 2014-01-22; First posted 2014-01-24 (Estimated); Last update posted 2018-06-21 (Actual); Status verified 2018-06

CONDITIONS: Stage 4 Pulmonary Sarcoidosis
Keywords: Sarcoidosis, pulmonary rehabilitation
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary rehabilitation (Experimental): Sarcoidosis patients will realize a pulmonary rehabilitation program
  Interventions: Other: Pulmonary rehabilitation program
- Controls (No Intervention): Sarcoidosis patients who do not achieve a respiratory rehabilitation program but will have physical activity counseling.

INTERVENTIONS:
Other: Pulmonary rehabilitation program — Pulmonary rehabilitation program should follow ATS/ERS Guidelines (2006)
  Arms: Pulmonary rehabilitation

SUMMARY:
The primary objective of the study is to assess the improvement of daily activity in subjects with Stage IV Pulmonary Sarcoidosis one year after the conduct of a pulmonary rehabilitation program.

The secondary objectives are the following:

* assess the improvement of daily activity at several times : 2, 6 and 12 months after the beginning of a pulmonary rehabilitation program
* assess the improvement of exercise capacity by tests used in medical practice
* assess the correlation between daily activity and exercise capacity
* assess the improvement of dyspnea
* assess the improvement of quality of life and psychological state

DETAILED DESCRIPTION:
The primary objective of the study is to assess the improvement of daily activity in subjects with Stage IV Pulmonary Sarcoidosis one year after the conduct of a pulmonary rehabilitation program

The secondary objectives are the following :

* assess the improvement of daily activity at several times : 2, 6 and 12 months after the beginning of a pulmonary rehabilitation program
* assess the improvement of exercise capacity by tests used in medical practice
* assess the correlation between daily activity and exercise capacity
* assess the improvement of dyspnea
* assess the improvement of quality of life and psychological state

ELIGIBILITY:
Inclusion Criteria:

* Stage IV Sarcoidosis
* No hospitalization for respiratory distress in the 3 months preceding the inclusion
* Dyspnea on exertion
* Age over 18 years

Exclusion Criteria:

* Physical disability does not allow the creation of a rehabilitation program
* Inability to give written consent to the study
* Refusal of contraception in women of childbearing age
* Inability to participate in the entire study
* No cover by the social security system
* Inability to perform self-questionnaires etude

The trial does not include special populations include:

* Pregnant women
* Breastfeeding women
* People in emergencies
* Persons unable to consent
* Persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-07-10 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Daily activity assessed by time (in minutes) spent in moderate activity (superior to 2,5 MET) | 12 months
  In everyday life, it corresponds to a walking in 5 km/h or in domestic chores. This measure will be realized by using Armband's accelerometer, in ambulatory. The measure will be realized over a period of 4 full days including the weekend.

SECONDARY OUTCOMES:
Daily activity assessed by time spent in moderate activity (superior to 2,5 MET) | 2 and 6 months
exercise capacity assessed by symptom-limited cardiopulmonary exercise test, 6 minutes walk test, endurance test on bicycle, St Etienne questionnaire, 6 minutes stepper test | 2, 6 and 12 months
MRC scale for dyspnea | 2, 6 and 12 months
Questionnaire to evaluate quality of life and/or psychological state : VSRQ | 2, 6 and 12 months
Questionnaire to evaluate quality of life and/or psychological state : MRF 28 | 2, 6 and 12 months
Questionnaire to evaluate quality of life and/or psychological state : HAD | 2, 6 and 12 months
Questionnaire to evaluate quality of life and/or psychological state : FAS | 2, 6 and 12 months
Questionnaire to evaluate quality of life and/or psychological state : DIRECT | 2, 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoît WALLAERT, MD PhD, Principal Investigator — Clinique des Maladies Respiratoires, CHRU de Lille; Frédéric BART, MD, Principal Investigator — Service de Pneumologie, CH Béthune; Dominique VALEYRE, MD PhD, Principal Investigator — Service de pneumologie, Hôpital Avicenne AP-HP; Dominique ISRAEL-BIET, MD PhD, Principal Investigator — Service de Pneumologie, Hôpital européen Georges Pompidou. AP-HP; Jean AMOURETTE, MD, Principal Investigator — Service de Pneumologie, CH Arras; Yves PACHECO, MD PhD, Principal Investigator — Centre Hospitalier Lyon Sud; Vincent COTTIN, MD PhD, Principal Investigator — Service de Pneumologie, Hôpital Louis Pradel, Lyon; Martine REYNAUD-GAUBERT, MD PhD, Principal Investigator — CHU Nord, APHM Marseille; Sylvie LEROY, MD, Principal Investigator — Service de Pneumologie, Hôpital Pasteur - Pavillon H, CHU de Nice; Gaëtan DESLEE, MD, Principal Investigator — Hôpital Maison Blanche, CHU de Reims; François STEENHOUWER, MD, Principal Investigator — Service de Pneumologie, Hôpital Victor Provo, Roubaix; Alain DIDIER, MD, Principal Investigator — Clinique des Voies Respiratoires, Hôpital Larrey, Toulouse
Locations (11):
- France (11):
  - Clinique des Maladies Respiratoires, CHRU de LILLE, Lille, Nord
  - Service de Pneumologie, CH Béthune, Béthune, Pas De Calais
  - Service de Pneumologie, CH Arras, Arras
  - Service de pneumologie, Hôpital Avicenne AP-HP, Bobigny
  - CHU Nord, APHM Marseille, Marseille
  - Service de Pneumologie, Hôpital Pasteur - Pavillon H, CHU de Nice, Nice
  - Service de Pneumologie, Hôpital européen Georges Pompidou. AP-HP, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Hôpital Maison Blanche, CHU de Reims, Reims
  - Service de Pneumologie, Hôpital Victor Provo, Roubaix
  - Clinique des Voies Respiratoires, Hôpital Larrey, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wallaert B, Kyheng M, Labreuche J, Stelianides S, Wemeau L, Grosbois JM. Long-term effects of pulmonary rehabilitation on daily life physical activity of patients with stage IV sarcoidosis: A randomized controlled trial. Respir Med Res. 2020 Mar;77:1-7. doi: 10.1016/j.resmer.2019.10.003. Epub 2019 Oct 28. PMID 31855785